CLINICAL TRIAL: NCT01706913
Title: A Randomized Controlled Study to Assess the Impact of Dermatology Consultations on the Hospital Course of Patients Admitted for Cellulitis
Brief Title: Study Assessing Impact of Dermatology Consultation for Patients Admitted With Cellulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dermatology Foundation (Other)
Responsible Party: Principal Investigator, Daniela Kroshinsky, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DermFound-2008A058574
Record Dates: First submitted 2012-09-25; First posted 2012-10-15 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No consult (No Intervention): Those who are in the control group will follow internal medicine hospitalist recommendations alone which will include when and what type of post-discharge follow-up appointments the patient will have. We would like to emphasize that as part of the standard of care, patients in the control arm may still receive a dermatology consult if it is deemed necessary and/or requested. We will not prevent patients or the patient's team of caregivers from requesting a dermatology consultation during the course of hospitalization. A follow-up phone call will be performed two weeks after discharge for patients in the control group in order to confirm the patient's outcome. There will also be a medical record review one month after the patient's initial discharge from the hospital to assess for readmission
- Dermatology Consult (Active Comparator): The patients randomized to the treatment group will obtain a dermatology evaluation within 24 hours of being admitted to MGH for their cellulitis. The skin and lymph node exam performed by the dermatologist on patients in the treatment group will be documented in the LMR for the subjects' medical records. Patients who are readmitted for cellulitis within one month of being discharged from the hospital will be considered treatment failures. Patients in the treatment group will have a follow-up visit in dermatology clinic within two weeks after being discharged. There will also be a medical record review performed one month after the patient's initial discharge from the hospital to assess for readmission.
  Interventions: Other: Dermatology consult

INTERVENTIONS:
Other: Dermatology consult
  Arms: Dermatology Consult

SUMMARY:
This is a randomized, controlled study to compare patients evaluated and managed by internal medicine hospitalists alone versus patients who are additionally evaluated by a dermatologist when they are admitted to the hospital, aiming to demonstrate that hospital admissions for cellulitis that involve early dermatology consultation will reduce hospital length of stay, readmission rates, prevalence of pseudocellulitis, cost, and antibiotic usage. The hypothesis of this study is that obtaining inpatient dermatology consultations, within 24 hours of a patient being admitted to the hospital for cellulitis, will reduce the length of stay, readmission rate, cost, and antibiotic usage of the patient"s admission as well as properly evaluate and diagnose patients with pseudocellulitis. The primary objective will be to measure the difference in the length of stay for patients who are randomized to a dermatology consultation within 24 hours of hospital admission (active arm) versus being managed by an internal medicine hospitalist alone, as is the standard of care (control arm). The length of stay for each arm will be assessed once the study has been completed. The secondary endpoint will be to measure readmission rates for cellulitis after patients are discharged from the hospital. An additional endpoint will be to determine if antibiotic usage differs between patients randomized to a dermatology consultation and those not. Exploratory analyses will assess the percentage of patients with a concomitant known predisposing factor for recurrent cellulitis such as lymphedema, leg ulceration, tinea pedis, or onychomycosis, as well as the association of fever >100.5 F and a history of a prior episode of cellulitis.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent
* Able to complete study and comply with study procedures
* Presumed clinical diagnosis of cellulitis by medicine team

Exclusion Criteria:

* Have a known postoperative site infection or abscess
* Have a human/animal bite
* Have known osteomyelitis
* Have a hardware/line infection
* Are under the age of 18
* Have a history of transplantation less than six months after initial transplant and/or if they have had an episode of acute rejection in the last 90 days
* Known use of antithymocyte globulin or campath in the last 6 months or more than 20 mg/day of prednisone for more than 30 days -
* Are a known prisoner.
* Are decisionally-impaired.
* Have abnormal vital signs defined as systolic blood pressure <90 mmHg, diastolic blood pressure <80 mmHg, heart rate greater than 90 beats per minute or less than 50 beats per minute, respiratory rate greater than 20, or temperature > 100.5 F.
* Are known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2012-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic usage | 2 weeks after discharge from hospital stay
  We will be measuring the difference between antibiotic usage in patients in the control group as compared with the treatment group

SECONDARY OUTCOMES:
Length of hospital stay | Will be measured at day of patient discharge
  We will be comparing the length of admission between the control group and the treatment group to assess whether a dermatology consult has any impact on the length of a patient's hospital stay.

OTHER OUTCOMES:
Readmission rate | 2 weeks after patient discharge
  We will be measuring the readmission rate among patients in both groups in order to discover whether a dermatology consult has an impact on readmission rates among patients with cellultis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Kroshinsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ko LN, Garza-Mayers AC, St John J, Strazzula L, Vedak P, Shah R, Dobry AS, Rao SR, Milne LW, Parry BA, Kroshinsky D. Effect of Dermatology Consultation on Outcomes for Patients With Presumed Cellulitis: A Randomized Clinical Trial. JAMA Dermatol. 2018 May 1;154(5):529-536. doi: 10.1001/jamadermatol.2017.6196. PMID 29453872